CLINICAL TRIAL: NCT00949780
Title: Use of Chloral Hydrate to Perform Auditory Brainstem Response (ABR)
Brief Title: Chloral Hydrate to Perform Auditory Brainstem Response (ABR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Mariana Lopes Favero, Pontificia Universidade Catolica de São Paulo
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PUCSP-HC
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Last update posted 2009-07-31 (Estimated); Status verified 2009-07

CONDITIONS: Auditory Brainstem Response in Children; Sedation With Chloral Hydrate
Keywords: ABR; Chloral Hydrate; Sedation; Children
MeSH Terms: interventions — Chloral Hydrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chloral hydrate , sedative (Active Comparator)
  Interventions: Drug: Chloral Hydrate

INTERVENTIONS:
Drug: Chloral Hydrate

SUMMARY:
Chloral Hydrate (CH) is a well known drug for sedative and hypnotic purposes used in pediatric and dental procedures owing to the low depressive effect it has over respiratory and cardiac systems. Despite that, the literature reports cases of heart arrhythmia and sudden death in children, especially when using high doses, probably due to accumulation of serum trichloroethanol, an intermediate metabolite resulting from the liver metabolism of the drug. A possible carcinogenic action observed in guinea pigs has also been reported, even though it has not been confirmed in human beings.

Among the least severe complications there are paradoxical agitation, nausea, vomiting and excessive sleepiness.

CH is the drug of choice to sedate children undergoing Auditory Brainstem Response test (ABR), in which any movement or muscle contraction may generate artifacts that interfere in the analysis.

Profound sleep that lasts on average one hour is rapidly induced depending on the used dose, causing no residual sleepiness after this period; however, there is consensus in the literature about the best dose, which may range from 40 to 100 mg/kg.

Objective:

To assess the efficacy of CH as a sedative agent in performing ABR in children and to systematize its use.

ELIGIBILITY:
Inclusion Criteria:

* no success in previous attempts to perform the test during natural sleep

Exclusion Criteria:

* severe heart or lung disease

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2007-10; Primary Completion 2008-03 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
36 patients slept | one hour

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Mariana Lopes Favero, São Paulo, São Paulo
  - Derdic-Pucsp, São Paulo, São Paulo